CLINICAL TRIAL: NCT04943861
Title: Exploring the Consequences of Food Insecurity and Harnessing the Power of Peer Navigation and mHealth to Reduce Food Insecurity and Cardiometabolic Comorbidities Among Persons With HIV
Brief Title: Human Immunodeficiency Virus (HIV) Food Insecurities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: University of North Carolina, Greensboro (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00075503; R01NR020307 (NIH)
Record Dates: First submitted 2021-06-22; First posted 2021-06-29 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Food Insecurities; Cardiometabolic Comorbidities; HIV; PreDiabetes; Type 2 Diabetes Mellitus (T2DM)
Keywords: Food Insecurity
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2 | interventions — Secure resin cement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- weCare/Secure (Active Comparator): The weCare intervention is based on the social cognitive and empowerment theories and social support and is currently designed to reduce missed HIV care appointments and increase viral suppression among PWH who are newly diagnosed or out of care through the use of peer navigation and mHealth
  Interventions: Behavioral: weCare/Secure
- Usual Care (Other): There is no peer navigation within usual care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: weCare/Secure — The weCare intervention is based on the social cognitive and empowerment theories and social support and is currently designed to reduce missed HIV care appointments and increase viral suppression among PWH who are newly diagnosed or out of care through the use of peer navigation and mHealth
  Arms: weCare/Secure
Other: Usual Care — There is no peer navigation within usual care.
  Arms: Usual Care

SUMMARY:
The objectives of this study are to better understand how FI (food insecurities) contributes to the development of cardiometabolic comorbidities among PWH (People with HIV) and to test a novel bilingual FI intervention designed to reduce these comorbidities among food insecure PWH. The PI and staff will conduct this study in partnership with the Wake Forest Infectious Diseases Specialty Clinic, one of the largest Ryan White-funded clinics in North Carolina, which serves more than 2,000 PWH annually from a predominantly rural catchment area that includes South Central Appalachia. This area has high rates of both FI and HIV.

DETAILED DESCRIPTION:
The proposed study the team has created a conceptually integrated, mixed methods study that includes

* Longitudinal data collection to explore the difference in the prevalence and incidence of cardiometabolic comorbidities between food secure and insecure PWH
* Implementation and evaluation of the weCare/Secure intervention designed to improve insulin sensitivity among food insecure PWH with prediabetes or Type 2 diabetes (T2DM)
* Semi-structured individual in-depth interviews to understand the effect of the intervention on FI and insulin sensitivity among participants in an randomized controlled trial (RCT) trial
* Broad dissemination of study findings to inform both research and clinical practice

ELIGIBILITY:
Inclusion Criteria:

* participant must be a patient of the Wake Forest Infectious Diseases Specialty Clinic
* be living with HIV
* ≥18 years of age
* provide informed consent

Exclusion Criteria:

* unable to speak English or Spanish
* have cognitive impairment that would prevent participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) scores | Baseline
  Healthy Range: 1.0 (0.5-1.4) - Less than 1.0 means you are insulin-sensitive which is optimal. Above 1.9 indicates early insulin resistance
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) scores | Month 12
  Healthy Range: 1.0 (0.5-1.4) - Less than 1.0 means you are insulin-sensitive which is optimal. Above 1.9 indicates early insulin resistance
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) scores | Month 24
  Healthy Range: 1.0 (0.5-1.4) - Less than 1.0 means you are insulin-sensitive which is optimal. Above 1.9 indicates early insulin resistance
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) scores | Month 36
  Healthy Range: 1.0 (0.5-1.4) - Less than 1.0 means you are insulin-sensitive which is optimal. Above 1.9 indicates early insulin resistance

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Rhodes, PhD, Principal Investigator — Wake Forest Health Sciences
Locations (1):
- Wake Forest Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Sharing data generated from this study is an essential part of our proposed activities. This study will generate both quantitative and qualitative data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Last 6 months of Year 5
Access Criteria: De-identified data and associated documentation (including codebooks) will be available from the Principal Investigators under a data-sharing agreement with users that provides for a commitment to:
  (1) using the data for research purposes; (2) securing the data using appropriate computer technology; and (3) to destroying or returning the data after analyses are completed

REFERENCES:
- [Derived] Tanner AE, Palakshappa D, Morse CG, Mann-Jackson L, Alonzo J, Garcia M, Wright E, Dharod A, Isom S, Sucaldito AD, Aviles LR, Rhodes SD. Exploring the consequences of food insecurity and harnessing the power of peer navigation and mHealth to reduce food insecurity and cardiometabolic comorbidities among persons with HIV: protocol for development and implementation trial of weCare/Secure. Trials. 2022 Dec 12;23(1):998. doi: 10.1186/s13063-022-06924-3. PMID 36510319